CLINICAL TRIAL: NCT03434028
Title: Crystalloid Liberal or Vasopressors Early Resuscitation in Sepsis
Acronym: CLOVERS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Boyd Taylor Thompson, PETAL CCC Prinicipal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PETAL03 CLOVERS
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Results first posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Septic Shock
Keywords: Fluid management; Sepsis-induced hypotension; vasopressors
MeSH Terms: conditions — Shock, Septic | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Restrictive Fluids (Other): The general approach will be to use vasopressors to treat hypotension as opposed to intravenous fluids. Maintenance fluids should not be used.
  Interventions: Drug: Early Vasopressors
- Liberal Fluids (Other): The general approach is to use fluid boluses to treat hypotension.
  Interventions: Other: Early Fluids

INTERVENTIONS:
Drug: Early Vasopressors — Norepinephrine will be used as preferred vasopressor and titrated to achieve mean arterial pressure (MAP) between 65 mmHg and 75 mmHg. "Rescue fluids" may be administered as 500ml boluses if predefined rescue criteria are met.
  Other Names: Norepinephrine
  Arms: Restrictive Fluids
Other: Early Fluids — Additional 2 liter intravenous fluid infusion upon enrollment (may forego second liter if MAP/SBP and heart rate are normalized and clinical assessment if patient is fluid replete after the first liter). Administer 500ml fluid boluses for fluid triggers until 5 liters administered or development of clinical signs of acute volume overload develop. "Rescue vasopressors" may be administered after 5 liters of fluid, for development of acute volume overload, or if other predefined rescue criteria are met. Any type of isotonic crystalloid (normal saline, ringers lactate, balanced solution such as plasmalyte) is permitted.
  Other Names: Balanced crystalloid solution
  Arms: Liberal Fluids

SUMMARY:
Multicenter, prospective, phase 3 randomized non-blinded interventional trial of fluid treatment strategies in the first 24 hours for patients with sepsis-induced hypotension. The aim of the study is to determine the impact of a restrictive fluids strategy (vasopressors first followed by rescue fluids) as compared to a liberal fluid strategy (fluids first followed by rescue vasopressors) on 90-day in-hospital mortality in patients with sepsis-induced hypotension.

DETAILED DESCRIPTION:
Primary Hypothesis: Restrictive (vs liberal) fluid treatment strategy during the first 24 hours of resuscitation for sepsis-induced hypotension will reduce 90-day in-hospital mortality.

1. We will emphasize early screening and protocol initiation, and enroll a maximum of 2320 patients with suspected sepsis-induced hypotension.

   * All patients will receive at least 1 liter of fluids prior to meeting study inclusion criteria (and no more than 3 liters prior to randomization).
   * Patients will be enrolled within 4 hours of meeting study inclusion criteria
   * Any type of isotonic crystalloid (normal saline, ringers lactate, or a balanced solution such as plasmalyte) is permitted.
2. Restrictive Fluids (Early Vasopressors) Group

   * Norepinephrine will be used as preferred vasopressor and titrated to achieve mean arterial pressure (MAP) between 65 mmHg and 75 mmHg
   * "Rescue fluids" may be administered as 500ml boluses if predefined rescue criteria are met
3. Liberal Fluids (Fluids First)

   * 2 liter infusion upon enrollment (may forego second liter if MAP/SBP and heart rate are normalized and clinical assessment if patient is fluid replete after the first liter).
   * Administer 500ml fluid boluses for fluid triggers until 5 liters administered or development of clinical signs of acute volume overload develop
   * "Rescue vasopressors" may be administered after 5 liters of fluid, for development of acute volume overload, or if other predefined rescue criteria are met

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* A suspected or confirmed infection (broadly defined by administration or planned administration of antibiotics)
* Sepsis-induced hypotension defined as systolic blood pressure < 100 mmHg or MAP < 65 mmHg after a minimum of at least 1 liter of fluid (*Fluids inclusive of pre-hospital fluids; blood pressure must be below any known or reported pre-morbid baseline).

Exclusion Criteria:

* More than 4 hours elapsed since meeting inclusion criteria or 24 hours elapsed since admission to the hospital
* Patient already received 3 liters of intravenous fluid (includes prehospital volumes)
* Unable to obtain informed consent
* Known pregnancy
* Hypotension suspected to be due to non-sepsis cause (e.g. hemorrhagic shock)
* Blood pressure is at known or reported baseline level
* Severe Volume Depletion from an acute condition other than sepsis. In the judgment of the treating physician, the patient has an acute condition other than sepsis causing (or indicative) of *severe volume depletion; Examples include: Diabetic ketoacidosis, high volume vomiting or diarrhea, hyperosmolar hyperglycemic state, and nonexertional hyperthermia (heat stroke); severe is defined by the need for substantial intravenous fluid administration as part of routine clinical care
* Pulmonary edema or clinical signs of new fluid overload (e.g. bilateral crackles, new oxygen requirement, new peripheral edema, fluid overload on chest x-ray)
* Treating physician unwilling to give additional fluids as directed by the liberal protocol
* Treating physician unwilling to use vasopressors as directed by the restrictive protocol.
* Current or imminent decision to withhold most/all life-sustaining treatment; this does not exclude those patients committed to full support except cardiopulmonary resuscitation
* Immediate surgical intervention planned such that study procedures could not be followed
* Prior enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1563 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Alan Schoenfeld, PhD, Principal Investigator — Massachusetts General Hospital
Locations (49):
- United States (49):
  - University of Arizona, Tucson, Arizona
  - UCSF Fresno, Fresno, California
  - Ronald Reagan UCLA, Los Angeles, California
  - UCSF San Francisco, San Francisco, California
  - Stanford University Hospital, Stanford, California
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - University Medical Center (LSU), New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - St. Vincent Hospital, Worcester, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mt. Sinai Hospital, New York, New York
  - Montefiore Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health and Science University OHSU, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC Mercy, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - University Virginia Medical Center, Charlottesville, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Swedish Hospital First Hill, Seattle, Washington

REFERENCES:
- [Derived] Oshima K, Yan B, Tao R, Amorim G, Di Gravio C, McMurtry SA, Burke RC, Nam Y, Nikolli I, Kravitz MS, Stephenson D, Issaian A, Hansen KC, D'Alessandro A, Douglas IS, Self WH, Lindsell CJ, Leroux C, Ringor A, Matthay MA, Schildcrout JS, Shapiro NI, Schmidt EP. Plasma chondroitin sulfate predicts the effectiveness of fluid resuscitation strategies in patients with sepsis. J Clin Invest. 2026 Feb 3:e202480. doi: 10.1172/JCI202480. Online ahead of print. PMID 41632536
- [Derived] Oshima K, Di Gravio C, Yan B, McMurtry SA, Burke R, Levoir LM, Kravitz MS, Stephenson D, Issaian A, Hansen KC, D'Alessandro A, Douglas IS, Self WH, Lindsell CJ, Schildcrout JS, Schmidt EP, Shapiro NI. Endothelial Glycocalyx Degradation in Sepsis: Analysis of the Crystalloid Liberal or Vasopressors Early Resuscitation in Sepsis (CLOVERS) Trial, a Multicenter, Phase 3, Randomized Trial. Ann Am Thorac Soc. 2025 Sep;22(9):1382-1393. doi: 10.1513/AnnalsATS.202501-012OC. PMID 40315385
- [Derived] Jorda A, Douglas IS, Staudinger T, Heinz G, Bergmann F, Oberbauer R, Sengolge G, Zeitlinger M, Jilma B, Shapiro NI, Gelbenegger G. Fluid management for sepsis-induced hypotension in patients with advanced chronic kidney disease: a secondary analysis of the CLOVERS trial. Crit Care. 2024 Jul 11;28(1):231. doi: 10.1186/s13054-024-05019-6. PMID 38992663
- [Derived] National Heart, Lung, and Blood Institute Prevention and Early Treatment of Acute Lung Injury Clinical Trials Network; Shapiro NI, Douglas IS, Brower RG, Brown SM, Exline MC, Ginde AA, Gong MN, Grissom CK, Hayden D, Hough CL, Huang W, Iwashyna TJ, Jones AE, Khan A, Lai P, Liu KD, Miller CD, Oldmixon K, Park PK, Rice TW, Ringwood N, Semler MW, Steingrub JS, Talmor D, Thompson BT, Yealy DM, Self WH. Early Restrictive or Liberal Fluid Management for Sepsis-Induced Hypotension. N Engl J Med. 2023 Feb 9;388(6):499-510. doi: 10.1056/NEJMoa2212663. Epub 2023 Jan 21. PMID 36688507
- [Derived] Self WH, Semler MW, Bellomo R, Brown SM, deBoisblanc BP, Exline MC, Ginde AA, Grissom CK, Janz DR, Jones AE, Liu KD, Macdonald SPJ, Miller CD, Park PK, Reineck LA, Rice TW, Steingrub JS, Talmor D, Yealy DM, Douglas IS, Shapiro NI; CLOVERS Protocol Committee and NHLBI Prevention and Early Treatment of Acute Lung Injury (PETAL) Network Investigators. Liberal Versus Restrictive Intravenous Fluid Therapy for Early Septic Shock: Rationale for a Randomized Trial. Ann Emerg Med. 2018 Oct;72(4):457-466. doi: 10.1016/j.annemergmed.2018.03.039. Epub 2018 May 10. PMID 29753517

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Restrictive Fluids | Liberal Fluids
Started | 782 | 781
Completed | 782 | 781
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Restrictive Fluids | Liberal Fluids | Total
Number analyzed (Participants) | 782 | 781 | 1563
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (16) | 59.9 (15.9) | 59.5 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 371 | 366 | 737
  Male | 411 | 415 | 826
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 4 | 12
  Asian | 26 | 26 | 52
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 134 | 112 | 246
  White | 532 | 570 | 1102
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 78 | 67 | 145
Region of Enrollment [Number; unit: participants]
  United States | 782 | 781 | 1563
Hispanic or Latino ethnic group [Count of Participants; unit: Participants]
  yes | 118 | 108 | 226
  no | 628 | 646 | 1274
  not reported | 36 | 27 | 63
Sequential Organ Failure Assessment (SOFA) score [Mean (Standard Deviation); unit: units on a scale] — Higher SOFA score = worse outcome.CLOVERS clinically significant organ failure: SOFA score 2 or more points higher than baseline. Total score ranges: 0(min)-4(max) Score: Coagulation(platelets x10³/µL: 0:>150; 1:</=150; 2:</=100; 3:</=50; 4:</=20. Liver(bilirubin, mg/dL): 0:<1.2; 1: 1.2-1.9; 3: 2.0-5.9; 3: 6.0-11.9; 4:>11.9. Cardiovascular(hypotension): 0:none; 1: MAP <70 mmHg; 2: Dop</=5 or dob (any dose); 3:dop>5, epi</=0.1, or norepi</=0.1; 4: Dop>15, epi>0.1, or norepi>0.1. Renal(creatinine, mg/dL or urine output,ml/d): 0:<1.2; 1: 1.2-1.9; 3: 2.0-3.4; 3: 3.5-4.9 or <500; 4:>4.9 or <200.
  units on a scale | 3.4 (2.8) | 3.5 (2.7) | 3.4 (2.7)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 93.2 (12) | 93.8 (12.2) | 93.5 (12.1)
Time from meeting eligibility to randomization [Median (Inter-Quartile Range); unit: minutes] — Median time from meeting trial eligibility criteria to randomization
  minutes | 61 [26 to 116] | 60 [25 to 117] | 61 [26 to 116]
Location at Randomization [Count of Participants; unit: Participants]
  Emergency Department | 729 | 708 | 1437
  ICU | 44 | 62 | 106
  Other | 9 | 11 | 20
Volume of fluid administered before randomization [Median (Inter-Quartile Range); unit: mililiters] | 2050 [1500 to 2457] | 2050 [1371 to 2442] | 2050 [1450 to 2450]
Coexisting Conditions [Count of Participants; unit: Participants]
  Diabetes: Yes | 222 | 224 | 446
  Diabetes: No | 555 | 549 | 1104
  Diabetes: No reported | 5 | 8 | 13
  Chronic heart failure: Yes | 99 | 79 | 178
  Chronic heart failure: No | 678 | 694 | 1372
  Chronic heart failure: No reported | 5 | 8 | 13
  end-stage renal disease treated with hemodialysis: Yes | 33 | 40 | 73
  end-stage renal disease treated with hemodialysis: No | 744 | 733 | 1477
  end-stage renal disease treated with hemodialysis: No reported | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Death Before Discharge Home by Day 90
Description: The primary outcome was death from any cause before discharge home by day 90. Point estimates were from Kaplan-Meier curves. There were 109 deaths and 5 patients with censored data the restrictive fluid group and 116 deaths and 4 patients with censored data in the liberal group. We defined home as the same setting or a setting similar to the one where the patient resided before becoming ill. Thus, if a patient originated from a private residence and was discharged from the hospital to a rehabilitation setting, we assessed for vital status until return to the private residence.Vital status was determined using any of the following methods: medical record review, phone calls to patient, proxy or healthcare facility, review of obituaries, or information from the Centers for Disease Control and Prevention's National Death Index (NDI).
Time Frame: From randomization to discharge home up to and including day 90.
Population: There were 109 deaths and 5 patients with censored data the restrictive fluid group. There were 116 deaths and 4 patients with censored data in the liberal group. Point estimates from the Kaplan-Meier curve.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Restrictive Fluids | Liberal Fluids
Number analyzed (Participants) | 782 | 781
percentage of participants | 14 [11.6 to 16.4] | 14.9 [12.4 to 17.4]
Statistical Analysis 1: Comparison: Restrictive Fluids vs Liberal Fluids; Test type: Superiority; p = 0.61, Z-test; difference in mortality rate = -0.9, 95% CI 2-sided [-4.4 to 2.6]

2. Secondary Outcome: Organ Support Free Days
Description: Defined as a patient being alive and without assisted breathing, new renal replacement therapy, or vasopressors (excluding vasopressor use prior to 48 hours). Any day that a patient is alive and without organ support will represent days alive and free of organ support.
Time Frame: 28 days after randomization
Population: We only report primary and secondary outcomes using available data without imputation. Because of missing data, the denominator may vary for selected outcomes as reported in the primary publication (PMID: 36688507).
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Restrictive Fluids | Liberal Fluids
Number analyzed (Participants) | 778 | 778
days | 24 [23.4 to 24.6] | 23.6 [23 to 24.3]
Statistical Analysis 1: Comparison: Restrictive Fluids vs Liberal Fluids; Test type: Superiority; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.5 to 1.2] — The mean values is an estimate from the Kaplan-Meier curve, thus it is correct as reported

3. Secondary Outcome: Ventilator Free Days (VFD)
Description: Ventilator-free days is defined to be 28 days minus the duration of mechanical ventilation through day 28. Participants who do not survive to day 28 are assigned zero ventilator-free days.
Time Frame: 28 days after randomization
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Restrictive Fluids | Liberal Fluids
Number analyzed (Participants) | 773 | 771
days | 23.4 [22.7 to 24.1] | 22.8 [22 to 23.5]
Statistical Analysis 1: Comparison: Restrictive Fluids vs Liberal Fluids; Test type: Superiority; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.4 to 1.6]

4. Secondary Outcome: Renal Replacement Free Days
Description: The number of calendar days between randomization and 28 days later that the patient is alive and without renal replacement therapy. Patients who died prior to day 28 are assigned zero renal replacement free days.
Time Frame: 28 days after randomization
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Restrictive Fluids | Liberal Fluids
Number analyzed (Participants) | 737 | 738
days | 24.1 [23.4 to 24.8] | 23.9 [23.2 to 24.6]
Statistical Analysis 1: Comparison: Restrictive Fluids vs Liberal Fluids; Test type: Superiority; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.8 to 1.2]

5. Secondary Outcome: Vasopressor Free Days
Description: The number of calendar days between day 2 (eligibility starting 48 hours post randomization) and 26 days later that the patient is alive and without the use of vasopressor therapy. Patients who died prior to day 28 are assigned zero vasopressor free days.
Time Frame: From study day 2 through day 28
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Restrictive Fluids | Liberal Fluids
Number analyzed (Participants) | 778 | 778
days | 22 [21.4 to 22.7] | 21.6 [20.9 to 22.3]
Statistical Analysis 1: Comparison: Restrictive Fluids vs Liberal Fluids; Test type: Superiority; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.5 to 1.3]

6. Secondary Outcome: ICU Free Days
Description: Defined as the number of days spent alive out of the ICU to day 28.
Time Frame: 28 days after randomization
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Restrictive Fluids | Liberal Fluids
Number analyzed (Participants) | 778 | 778
days | 22.8 [22.2 to 23.4] | 22.7 [22 to 23.3]
Statistical Analysis 1: Comparison: Restrictive Fluids vs Liberal Fluids; Test type: Superiority; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.8 to 1.0]

7. Secondary Outcome: Hospital Free Days to Discharge Home
Description: Days alive post hospital discharge through day 28. Patients who die on or prior to day 28 are assigned zero hospital free days.
Time Frame: 28 days after randomization
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Restrictive Fluids | Liberal Fluids
Number analyzed (Participants) | 778 | 778
days | 16.2 [15.4 to 17] | 15.4 [14.6 to 16.2]
Statistical Analysis 1: Comparison: Restrictive Fluids vs Liberal Fluids; Test type: Superiority; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-0.3 to 1.9]

8. Secondary Outcome: New Intubation With Invasive Mechanical Ventilation by 28 Days
Description: Patients who receive invasive mechanical ventilation via endotracheal or tracheostomy tube, except those intubated solely for a procedure and extubated within 24 hours, through to study day 28 meet this endpoint. Non-invasive mechanical ventilation will not be included as an outcome. This is a binary outcome.
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive Fluids | Liberal Fluids
Number analyzed (Participants) | 701 | 687
Participants | 77 | 87
Statistical Analysis 1: Comparison: Restrictive Fluids vs Liberal Fluids; Test type: Superiority; Risk Difference (RD) = -1.7, 95% CI 2-sided [-5.1 to 1.7]

9. Secondary Outcome: Initiation of Renal Replacement Therapy
Description: Patients receiving (new) renal replacement therapy through day 28. Patients with chronic renal replacement therapy initiated prior to the current sepsis illness were not eligible to meet this endpoint.
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive Fluids | Liberal Fluids
Number analyzed (Participants) | 738 | 738
Participants | 24 | 24
Statistical Analysis 1: Comparison: Restrictive Fluids vs Liberal Fluids; Test type: Superiority; Risk Difference (RD) = 0.0, 95% CI 2-sided [-1.8 to 1.8]

10. Secondary Outcome: Kidney Disease: Change in Creatinine-based Global Outcomes (KIDGO) Score Between Baseline and 72 Hours
Description: Assessment of renal function using the KDIGO staging system (using serum creatinine criteria only) between baseline and 72 hours post randomization to assess for de novo acute kidney injury (AKI) (e.g., meeting criteria for AKI by KDIGO criteria) or worsening AKI (e.g., increasing severity). Patients on chronic renal replacement therapy were not eligible for this endpoint determination.
  Scoring of 1-3 (using serum creatinine levels; a higher score indicates worsening kidney function):
  1. creatinine level 1.5-1.9 times baseline OR >/= 0.3 mg/dl (>/= 25.5 umol/l) increase
  2. creatinine level 2.0-2.9 times baseline
  3. creatinine level 3.0 times baseline OR increase in serum creatinine to >/=4.0mg/dl (>/= 353 umol/l) OR initiation of renal replacement therapy
Time Frame: 72 hours after randomization
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Restrictive Fluids | Liberal Fluids
Number analyzed (Participants) | 585 | 604
score on a scale | 0.35 [0.28 to 0.41] | 0.34 [0.28 to 0.41]
Statistical Analysis 1: Comparison: Restrictive Fluids vs Liberal Fluids; Test type: Superiority; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.1 to 0.1]

11. Secondary Outcome: Change in SOFA (Sepsis Related Organ Failure Assessment) Score
Description: SOFA score was calculated at enrollment and at 72 hours using clinically available data.Total score: 0-4 points; 4 = worst outcome. Values not available at baseline were assumed normal. 72 hours assessment: Closest previously known value was carried forward for missing values. SOFA Scoring Breakout (lower scores mean a better outcome; clinically significant organ failure for CLOVERS was defined as a SOFA score 2 or more points higher than baseline):
  * Coagulation( Platelets, ×10³/µL): Score = 0: >150; 1: </= 150; 2: </= 100; 3: </= 50; 4: </= 2
  * Liver (Bilirubin, mg/dL): Score: 0: <1.2; 1: 1.2-1.9; 2: 2.0-5.9; 3: 6.0-11.9; 4: >11.9
  * Cardiovascular(Hypotension): Score: 0: no hypotension; 1: Mean arterial pressure <70 mmHg; 2: Dopamine</=5 OR any dobutamine; 3: Dopanime >5, epinephrine </=0, or Norepi </=0.1; 4: Dop >15, epi >0.1, or norepi >0.1
  * Renal (Creatinine, mg/dL or urine output, ml/d): Score: 0: <1.2; 1: 1.2-1.9; 3: 2.0-3.4; 3: 3.5-4.9 or <500; 4: >4.9 or <200
Time Frame: 72 hours after randomization
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Restrictive Fluids | Liberal Fluids
Number analyzed (Participants) | 619 | 634
score on a scale | -0.7 [-0.9 to -0.4] | -0.8 [-1 to -0.5]
Statistical Analysis 1: Comparison: Restrictive Fluids vs Liberal Fluids; Test type: Superiority; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.4]

12. Secondary Outcome: Development of ARDS
Description: Presence and severity of ARDS is determined using the PaO2/FiO2 ratio or SpO2/FiO2 ratio and confirmation of ARDS through chest x-ray reviews.
Time Frame: 7 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive Fluids | Liberal Fluids
Number analyzed (Participants) | 757 | 758
Participants | 19 | 20
Statistical Analysis 1: Comparison: Restrictive Fluids vs Liberal Fluids; Test type: Superiority; Risk Difference (RD) = -0.1, 95% CI 2-sided [-1.7 to 1.5]

13. Secondary Outcome: New Onset Atrial or Ventricular Arrhythmia
Description: The occurrence of one or more episodes (sustained for more than 1 minute for SVT and AF, > 15 seconds for VT) during through day 28 will be recorded.
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive Fluids | Liberal Fluids
Number analyzed (Participants) | 779 | 778
Participants | 59 | 67
Statistical Analysis 1: Comparison: Restrictive Fluids vs Liberal Fluids; Test type: Superiority; Risk Difference (RD) = -1.0, 95% CI 2-sided [-3.7 to 1.7]

14. Secondary Outcome: Death From Any Cause at Any Location by Day 90
Description: Subjects were contacted at day 90 to ascertain their survival status via telephone contact with the patient or family members or by a review of medical records and publicly available data sources.
Time Frame: From randomization to and including day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive Fluids | Liberal Fluids
Number analyzed (Participants) | 768 | 773
Participants | 172 | 169
Statistical Analysis 1: Comparison: Restrictive Fluids vs Liberal Fluids; Test type: Superiority; Risk Difference (RD) = 0.5, 95% CI 2-sided [-3.6 to 4.7]

ADVERSE EVENTS:
Time Frame: Assessment for adverse events was performed from trial enrollment through study day 6 (five days after completion of the study fluid protocol) or Hospital discharge, whichever occurs first. All-Cause All-Location Mortality was assessed up to 90 days from randomization. Please note that this outcome measure differs from the primary outcome of death before discharge home by day 90 and includes deaths after discharge home before day 90.
Description: Events that were assessed to be serious or non-serious and that were considered to be related to study procedures or of uncertain relationship were captured. As noted previously, because of missing data the denominator may vary for selected outcomes. The number of patients at risk for adverse events is all patients randomized (no missing data). All deaths due to any cause to day 90 are reported.
Arm/Group | Restrictive Fluids | Liberal Fluids
All-Cause Mortality (participants affected / at risk) | 172/768 | 169/773
Serious Adverse Events (participants affected / at risk) | 18/782 | 19/781
Other Adverse Events (participants affected / at risk) | 4/782 | 14/781
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Restrictive Fluids (N=782) | Liberal Fluids (N=781)
Anemia (Blood and lymphatic system disorders) | 1 | 0 — Definitely not study related
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 — Definitely not study related
Cardiac Arrest (Cardiac disorders) | 1 | 0 — Definitely not study related
Polymorphic Vt (Cardiac disorders) | 1 | 0 — Probably not study related
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 — Probably or possibly study related
Gastrointestinal Bleeding (Gastrointestinal disorders) | 2 | 0 — Definitely not study related
Death (General disorders) | 1 | 0 — Probably not study related
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0 — Definitely not study related
Cholangitis (Hepatobiliary disorders) | 1 | 0 — Definitely not study related
Pneumonia (Infections and infestations) | 1 | 0 — Definitely not study related
Septic Shock (Infections and infestations) | 1 | 0 — Probably not study related
Lactic Acidosis (Metabolism and nutrition disorders) | 1 | 0 — Probably not study related
Cerebral Infarct (Nervous system disorders) | 1 | 0 — Probably not study related
Seizure (Nervous system disorders) | 1 | 0 — Definitely not study related
Hematuria (Renal and urinary disorders) | 1 | 0 — Definitely not study related
Worsening Kidney Failure (Renal and urinary disorders) | 1 | 0 — Probably not study related
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Probably not study related
Hypotension (Vascular disorders) | 1 | 0 — Definitely not study related
Peripheral Ischemia (Vascular disorders) | 2 | 0 — Probably or possibly study related/ Probably not study related
Cardiac Arrest (Cardiac disorders) | 0 | 2 — Definitely not study related
Pulmonary Edema (Cardiac disorders) | 0 | 2 — Probably or possibly study related
Flash Pulmonary Edema (Cardiac disorders) | 0 | 1 — Probably not study related
Fluid Overload (Cardiac disorders) | 0 | 3 — Probably not study related/Probably or possibly study related
Myocardial Ischemia, Elevated Troponin (Cardiac disorders) | 0 | 1 — Probably not study related
Tachycardia (Cardiac disorders) | 0 | 1 — Probably not study related
Death (General disorders) | 0 | 4 — Definitely not study related
Readmit (General disorders) | 0 | 1 — Definitely not study related
Cellulitis (Infections and infestations) | 0 | 1 — Probably not study related
Sepsis (Infections and infestations) | 0 | 2 — Probably not study related
Blisters (Skin and subcutaneous tissue disorders) | 0 | 1 — Probably not study related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Restrictive Fluids (N=782) | Liberal Fluids (N=781)
Chest Pain (Cardiac disorders) | 1 | 0 — Probably or possibly study related
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 — Probably or possibly study related
Seizure Vs Syncope Vasovagal (Nervous system disorders) | 1 | 0 — Probably not study related
Thrombosis Venous Deep (Vascular disorders) | 1 | 0 — Definitely not study related
Anemia (Blood and lymphatic system disorders) | 0 | 2 — Probably or possibly study related
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 — Definitely not study related
Bradycardia (Cardiac disorders) | 0 | 1 — Probably not study related
Fluid Overload (Cardiac disorders) | 0 | 3 — Probably or possibly study related/Probably not study related
Pulmonary Edema (Cardiac disorders) | 0 | 1 — Probably or possibly study related
Transfusion Associated Circulatory Overload (Cardiac disorders) | 0 | 1 — Probably or possibly study related
Renal Calculus (Renal and urinary disorders) | 0 | 1 — Definitely not study related
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Probably or possibly study related
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Probably or possibly study related
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Probably or possibly study related
Worsening Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Probably or possibly study related

LIMITATIONS AND CAVEATS:
All cause mortality: To clarify, we did not classify death as anticipated or not anticipated; nor did we collect cause of death for this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT03434028/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT03434028/SAP_001.pdf
  • Informed Consent Form (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT03434028/ICF_002.pdf